CLINICAL TRIAL: NCT02900391
Title: Urgent Care for the Elderly: Impairment and Home Care Services
Acronym: EPIGER
Status: Completed | Type: Observational
Sponsor: European Georges Pompidou Hospital (Other)
Responsible Party: Principal Investigator, Anne-Laure Feral-Pierssens, MD, European Georges Pompidou Hospital
Other Study IDs: EPIGER
Record Dates: First submitted 2016-09-01; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Impaired

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Elderly population is increasing quickly and their need for health care ressources through emergency care is also growing. While these patients are ageing physical impairment often happens along the way. Apart from senior homes, different types and levels of home care services have been developped in order to overcome or to adapt to these situations.

Our goals are:

* to assess mortality rate depending on home care services level for the elderly population consulting in the ED or being taken in charge by the Emergency Medical System in France.
* to describe this population in terms of autonomy, impairment and home care services

ELIGIBILITY:
Inclusion Criteria:

* patients aged 80 and over

Exclusion Criteria:

* aged<80 years old

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients aged 80 and over visiting the ED, taking in charge by SMUR (medical EMS) or calling SAMU (medical call center) during 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Actual)
Dates: Start 2016-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Mortality rate at hospital discharge | At hospital discharge or 30 days at most
  Mortality rate at hospital discharge

SECONDARY OUTCOMES:
Admission rate | Admission is decided on the first 24 hours after EMS or ED care, the day of the inclusion
  Admission in a medical, surgical or psychiatric unit are considered
Level of home care services | Questionnaires given the day of the inclusion
  Different items in a questionnaire are asked to the patient or family concerning weekly home care services use for patient usually (which type and how often)
Level of health care ressources | During the ED visit (less than 24 hours), the day of the inclusion
  Lab investigations, radiology, surgery, treatment administered

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feral-Pierssens AL, Toury G, Sehimi F, Peschanski N, Laribi S, Carpentier A, Kraif M, Carbonnier C, Duchateau FX, Freund Y, Juvin P; EPIGER IRU-SFMU study group. Emergency department outcome of elderly patients assisted by professional home services, the EPIGER study. BMC Geriatr. 2020 Sep 21;20(1):355. doi: 10.1186/s12877-020-01742-1. PMID 32957921